CLINICAL TRIAL: NCT06355141
Title: Investigation of Oral Structural and Functional Problems in Children With Autism Secondary IDs:
Brief Title: Oral Structural and Functional Problems in Children With Autism
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Kübra Şahan, Principal investigator, Hacettepe University
Other Study IDs: E-15189967-050.04-494458
Record Dates: First submitted 2024-03-09; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder; Chewing Problem; Drooling
Keywords: autism; chewing; drooling
MeSH Terms: conditions — Autism Spectrum Disorder; Sialorrhea; Autistic Disorder | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: oral assessment — observational oral assessment

SUMMARY:
This study aims to examine oral structural and functional problems in children with autism.

DETAILED DESCRIPTION:
In this descriptive study, children with autism will be screened for oral structural and functional problems. In this context, observational evaluation will be made. The presence of tongue thrust reflex, chewing performance and salivation control in children will be examined.Within the scope of the research, demographic data, parameters related to the oral motor development stage (time to transition to solid food and solid food, time to first teething) will be recorded according to parental report. Oral structural evaluation, including open mouth, high palate, oral hygiene and malocclusion, will be made observationally and recorded as present/absent. Within the scope of oral functional evaluation, tongue thrust reflex, chewing function and salivation control (dooling) will be evaluated.

The questions the investigators will test for this purpors; Q1:What oral structural and functional problems are seen in children with autism? Q2:What is the frequency of oral structural and functional problems seen in children with autism?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with autism,
* Not having any additional diagnosis other than autism,
* Age between 5-15 yers

Exclusion Criteria:

* Not being able to receive the commands required to obtain working data.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with autism (CwA) are five times more likely to experience feeding-related problems than their typically developing peers. Oral functional problems (chewing disorder, drooling of saliva), food selectivity, inappropriate mealtime interaction, abnormal eating speed (holding food in the mouth for a long time or fast feeding) and failure to eat the usual family diet are feeding-related reported in CwA.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-04-11 (Estimated); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-08-12 (Estimated)

PRIMARY OUTCOMES:
Demographic Information Form | 1 month
  Descriptive information will be recorded.
Time to achieve Oromotor skills | 1 month
  Parameters related to oromotor skills (transition time to additional food and solid food, initial teething time) were recorded based on a parental report.
Oral structural assessment | 1 month
  Oral structural evaluation, including open mouth, high-arched palate, oral hygiene and malocclusion, will be made observationally and recorded as present/absent. Evaluation of malocclusion will be made observationally while at rest. It will be recorded as normal, over jet, open bite, deep bite and cross bite present/absent.

SECONDARY OUTCOMES:
Chewing evaluation | 1 month
  Chewing function will be evaluated with the "Mastication Function Observation and Evaluation Tool (MOE, The Mastication Observation and Evaluation)". This tool includes an objective assessment of the chewing process in children. The child is monitored while eating a standard biscuit, and the observer scores the child's chewing skills based on 8 parameters. This assessment tool evaluates tongue movements, jaw movements, chewing time, food/saliva overflow, swallowing and coordination during chewing.
Drooling of saliva evaluation | 1 month
  Drooling frequency and sverity scale (DFSS) will be used. Drooling severity is scored between 1 and 5. It is scored as 1 meaning no saliva and dry, and 5 meaning continuous flow to the body and objects. Frequency is scored between 1 and 4. 1 means no drooling, 4 means constantly drooling.
Tongue thrust evaluation | 1 month
  The presence and severity of the tongue thrust will be evaluated with the Tongue ThrustRating Scale (TTRS). It evaluates the tongue thrust between 0 and 3 points. While 0 indicates that there is no tongue reflex, 3 indicates that the tongue is positioned outside the mouth, that is, a severe tongue thrust.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Kübra Söyler, Principal Investigator — Aydin Adnan Menderes University

IPD SHARING:
Plan to Share IPD: Undecided